CLINICAL TRIAL: NCT01300975
Title: Short Course of Intralesional Antimony for Bolivian Cutaneous Leishmaniasis
Brief Title: Intralesional Antimony for Bolivian Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Nacional de Dermatologia (Other)
Collaborators: The Alfred Berman Foundation for Medical Research (Unknown); Universidad Mayor de San Simón (Other); Hospital Dermatológico de Jorochito (Unknown); Proyecto OSCAR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABF-BO-2010-101
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2018-07

CONDITIONS: Leishmaniasis; Cutaneous Leishmaniasis
Keywords: Leishmaniasis; intralesional antimony; cryotherapy
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Cutaneous | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intralesional antimony (Experimental): 3 intralesional injections of antimony at D1, D3 and D7
  Interventions: Drug: pentavalent antimony
- Cryotherapy (Active Comparator): Liquid nitrogen until freezing at DF1 and D14
  Interventions: Procedure: cryotherapy
- Topical cream (Placebo Comparator): topical treatment 3 times a day during 21 days with an emollient cream
  Interventions: Drug: placebo cream

INTERVENTIONS:
Drug: pentavalent antimony — 3 intralesional injections of antimony at D1, D3 and D7
  Arms: Intralesional antimony
Procedure: cryotherapy — Frozing of lesions with liquid nitrogen ad D1 and D14
  Arms: Cryotherapy
Drug: placebo cream — topical emollient crean 3 times a day during 21 days
  Arms: Topical cream

SUMMARY:
Intralesional injection of antimony has been used for L major from Iran with a modest cure rate [56%: Asilian 2004]. However, this therapeutic approach has been used for L braziliensis from Brazil, with an attractive cure rate after 3 months of 80% [Oliveira-Neto 1997]. Because intralesional Sb injections is the local therapy with the best reported cure rate for South American L braziliensis disease, the species that causes disease in Bolivia, this pilot study of local therapy for bolivian L braziliensis disease will evaluate intralesional Sb therapy.

DETAILED DESCRIPTION:
Cutaneous leishmaniasis is endemic in the New World from approximately the US-Mexican border through Central America and the Northern part of South America down to the level of Rio de Janeiro.

Until recently, the standard treatment for the leishmaniases was pentavalent antimony (Glucantime or Pentostam). The cure rate for L panamensis in Colombia is 91%-93% [Soto, 1993; Velez, 1997], a large study with several formulations of antimony found a combined Bolivia-Colombia cure rate of 86% [Soto, 2004b], and the cure rate in Palos Blancos, Bolivia is 15 of 16 = 94% [ Soto, 2008]. Nevertheless, pentavalent antimonials have the disadvantages of multiple injections during at least 3 weeks and mild-moderate clinical toxicity: local pain at the site of injections and generalized myalgias and arthralgias that can be severe and responsible for partial or definitive interruption of therapy, gastrointestinal complaints, liver enzyme elevations, pancreatic enzyme elevations and more rarely but with danger for life ventricular repolarization problems [Soto, 2005, Velez 2010], all of which are particularly unpleasant for a localized moderate clinical problem such as cutaneous leishmaniasis that usually is not dangerous for the patient.

The oral agent Miltefosine has now been shown to be as effective as antimony in Colombia and Bolivia. In Colombia, the cure rate for miltefosine was 91% [Soto 2004a] and in the just-completed trial in Palos Blancos, the cure rate for miltefosine was 32 of 37 = 88 % . Side effects seen in patients with cutaneous disease that can be specifically attributed to the drug are nausea and vomiting of mild grade in approximately 25% of patients, and low-grade elevation of creatinine also in approximately 25% of patients [Soto 2001; Soto 2004]. Now that cutaneous leishmaniasis is affecting more women at reproductive age, there is a crucial inconvenient because miltefosine can't be taken during pregnancy and breastfeeding; additionally prolonged courses (4 weeks) makes more difficult adherence to therapy and emerge the risk of incomplete treatments or it might be necessary supervised administration during the full course.

For small, single lesions, the side effects and cost of systemic therapy with antimony or miltefosine may outweigh the advantage of cure. For such lesions, targeted local therapy would be attractive if it is effective. The cost of goods will be low, and systemic adverse events would be non-existent.

For these reasons, topical treatment of the leishmaniases is presently the subject of intense worldwide interest, including at a recent [July 2010] PAHO meeting in Colombia. The leading candidates are topical formulations of paromomyin, local heat since cutaneous leishmania are heat-sensitive, local freezing as per any dermatologic lesion, and intralesional injections of antimony. The ability of topical formulations of paromomycin to cure depends on penetration of this divalent cation into the lesion and thus depends on the precise formula for the cream in which the paromomycin is dissolved. Other than the combination of paromomycin plus MBCL in Vaseline, which had minimal efficacy in Colombia [Soto 1998], patented paromomycin-containing creams are under investigation but cannot be obtained except from Pharma. Reports of local thermotherapy have been published, but again the key issue is penetration of the agent [in this case, heat] to the lesion and the best approach is difficult to utilize because it requires a $25,000 machine and exists a risk of infections via electrodes.

Intralesional injection of antimony has also been used for L major from Iran, and also with a modest cure rate [56%: Asilian 2004]. However, this therapeutic approach has been used for L braziliensis from Brazil, with an attractive cure rate after 3 months of 80% [Oliveira-Neto 1997]. Because intralesional Sb injections is the local therapy with the best reported cure rate for South American L braziliensis disease, the species that causes disease in Bolivia, this pilot study of local therapy for bolivian L braziliensis disease will evaluate intralesional Sb therapy.

Cryotherapy has been used as sole therapy for L major from Iran. The cure rate was modest: 50-60% [Asilian 2004; Layegh 2009]. Nevertheless, cryotherapy may have an attractive cure rate against L braziliensis. Therefore, cryotherapy will also be evaluated in this pilot study.

Patients receiving intralesional Sb will be randomized vs vs patients receiving cryotherapy and also vs patients receiving an emollient cream Because Il Sb has perhaps more promise than cryotherapy, more patients will receive Il Sb (30) than will receive cryotherapy (20) The emollient cream may improve host response to the trauma of the parasitic process, nevertheless, emollient cream is a placebo treatment in the specifically antiparasitic sense. The spontaneous rate of cure is unknown in Bolivia, thus this group will serve to establish this key value and permit comparison of the IL Sb rate and the cryotherapy rate to it. Although 20 patients will be randomized to the "placebo" group, stopping rules are such that if 4 early patients or 6 total patients in this group fail, no further "placebo" patients will be entered into the trial.

ELIGIBILITY:
INCLUSION CRITERIA:

* Gender: Male or female
* Age: >12 yrs of age
* Clinicla presentation: 1-2 ulcerative lesions, each < 30 mm in largest diameter, and with a total lesion area <900 mm2.
* Parasitological confirmation of the lesion will be made by visualization or culture of leishmania from the biopsy or aspirate of the lesion.

EXCLUSION CRITERIA:

* Previous treatment for leishmaniasis: therapy with Sb, pentamidine, amphotericin B, miltefosine, imidazoles or allopurinol in the last 3 months
* Concomitant diseases by history that would be likely in the PI's opinion to interact, either positively or negatively, with IL Sb treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Complete clinical cure | six months
  100% epithelization, complete resolution of swelling and infiltration

SECONDARY OUTCOMES:
EKG changes associated with IL Sb, local reactions to cream and Cryo | six months
  Ealuation of clinical findings and changes in OKG, lipase and SGOT in patients receiving intralesional antimony

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berman, MD PhD, Study Chair — ABF; Jaime Soto, MD, Study Director — Fundacion Nacional de Dermatologia; Ernesto Rojas, MD, Principal Investigator — Universidad Mayor de San Simón
Locations (2):
- Bolivia (2):
  - CUNETROP - Universidad Mayor de San Simon, Cochabamba, CB
  - Hospital Dermatologico de Jorochito, Jorochito, SC

REFERENCES:
- [Background] Chaabane H, Masmoudi A, Dammak A, Kchaou W, Akrout F, Zribi M, Boudaya S, Turki H. [Cryotherapy with or without intralesional antimony in the treatment of cutaneous leishmaniasis]. Ann Dermatol Venereol. 2009 Mar;136(3):278-9. doi: 10.1016/j.annder.2008.09.016. Epub 2008 Dec 3. No abstract available. French. PMID 19328314
- [Result] Ranawaka RR, Weerakoon HS. Randomized, double-blind, comparative clinical trial on the efficacy and safety of intralesional sodium stibogluconate and intralesional 7% hypertonic sodium chloride against cutaneous leishmaniasis caused by L. donovani. J Dermatolog Treat. 2010 Sep;21(5):286-93. doi: 10.3109/09546630903287445. PMID 20438389
- [Derived] Soto J, Rojas E, Guzman M, Verduguez A, Nena W, Maldonado M, Cruz M, Gracia L, Villarroel D, Alavi I, Toledo J, Berman J. Intralesional antimony for single lesions of bolivian cutaneous leishmaniasis. Clin Infect Dis. 2013 May;56(9):1255-60. doi: 10.1093/cid/cit049. Epub 2013 Feb 6. PMID 23390069